CLINICAL TRIAL: NCT04561973
Title: Pain in Patients With Cystic Fibrosis in Rouen University Hospital
Acronym: MUCODOL
Status: Completed | Type: Observational
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Other Study IDs: 2019/318/OB
Record Dates: First submitted 2020-09-14; First posted 2020-09-24 (Actual); Last update posted 2022-02-21 (Actual); Status verified 2021-05

CONDITIONS: Pain; Cystic Fibrosis
Keywords: pain; cystic fibrosis; epidemiology; adults; children
MeSH Terms: conditions — Pain; Cystic Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: numerical rating scale — Patients seen for routine planned visits complete a self-administered retrospective questionnaire about pain during the last 3 months, and a prospective diary during the two weeks following the visit.

SUMMARY:
Objectif Principal

- To evaluate the intensity and frequency of pain episodes in patients with cystic fibrosis followed at the cystic fibrosis center of Rouen University Hospital, Normandy, France.

Objectifs secondaires

* To assess the relationship between pain and disease severity.
* To assess the relationship between pain and the age of the patient.
* To describe the pain locations.
* To describe the use of pharmacological or nonpharmacological treatment.
* To evaluate the procedural pain.

DETAILED DESCRIPTION:
Patients seen for routine planned visits complete a self-administered retrospective questionnaire about pain during the last 3 months, and a prospective diary during the two weeks following the visit.

Primary evaluation criteria :

Intensity and frequency of pain are evaluated with the prospective diary.

* The pain intensity is assessed by validated scales adapted to the patient's age (scale ranging from 0 to 10).

  0 to 6 years : numerical rating scale assessed by the parents. 4 to 7 years : Faces Pain Scale Revised. Children 6 years and older, adolescents and adults: numerical rating scale self-reported
* The pain frequency is completed twice a day (morning and evening) on the prospective pain diary.

Secondary evaluation criteria

* The disease severity, estimated using recent forced expiratory volume in one second (FEV1) (best measurement of the year before bronchodilator, collected in the patient's medical record)
* Pain locations, pharmacological or nonpharmacological treatment and procedural pain are evaluated using the diary and the questionnaire.
* Demographic data and characteristics of cystic fibrosis are collected using the medical file.

ELIGIBILITY:
Inclusion Criteria:

* Children and adults followed at the cystic fibrosis center of Rouen University Hospital, Normandy, France.
* Seen for routine planned visits.
* Having expressed their non-opposition or whose non-opposition was expressed by the parents or legal representatives for minors

Exclusion Criteria:

* Patients seen for an acute episode or exacerbation outside of routine planned visits or patient hospitalized.
* Major patient under legal protection.
* Major patient having problems understanding the oral and written French language or child whose parents or legal representatives have problems understanding the oral and written French language.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Children and adults followed at the cystic fibrosis center of Rouen University Hospital, Normandy, France
Sampling Method: Non-Probability Sample
Enrollment: 109 (Actual)
Dates: Start 2019-11-04 (Actual); Primary Completion 2020-10-15 (Actual); Study Completion 2020-11-01 (Actual)

PRIMARY OUTCOMES:
To evaluate the intensity and frequency of pain episodes in patients with cystic fibrosis followed at the cystic fibrosis center of Rouen University Hospital, Normandy, France | 14 days
  Intensity and frequency of pain are evaluated with the prospective diary. The pain intensity is assessed by validated scales adapted to the patient's age (scale ranging from 0 to 10).
  0 to 6 years : numerical rating scale assessed by the parents. 4 to 7 years : Faces Pain Scale Revised. Children 6 years and older, adolescents and adults: numerical rating scale self-reported The pain frequency is completed twice a day (morning and evening) on the prospective pain diary.

SECONDARY OUTCOMES:
To assess the correlation between pain and disease severity | 14 days
  The disease severity is estimated using recent forced expiratory volume in one second (FEV1) (best measurement of the year before bronchodilator), collected in the patient's medical record. The correlation between pain and the disease severity will be studied with a Spearman's correlation coefficient.
To assess the correlation between pain and the age of the patient. | 14 days
  Age of the patient is collected using the medical file. The correlation between pain and the age will be studied with a Spearman's correlation coefficient.
To describe the pain locations. | 14 days
  Pain locations are evaluated using the prospective diary and the self-administered retrospective questionnaire.
To describe the use of pharmacological or nonpharmacological treatment. | 14 days
  The pharmacological or nonpharmacological treatments are evaluated using the prospective diary (did you take a treatment for that pain episode ?) and the self-administered retrospective questionnaire. The efficacity of the treatment is evaluated with the diary (relief or not) et the questionnaire (Likert-type rating scale : Always, often, rarely, never).
To evaluate the procedural pain. | 3 months
  The procedural pain and the proposed pain treatment are evaluated using the self-administered retrospective questionnaire.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU, Rouen, Nomandie, France